CLINICAL TRIAL: NCT03666091
Title: Etude et Suivi Des POlyarthrites Indifférenciées Récentes
Brief Title: Study and Monitoring of Early Undifferentiated Arthritis
Acronym: ESPOIR
Status: Completed | Type: Observational
Sponsor: Societe Francaise de Rhumatologie (Other)
Collaborators: Amiens University Hospital (Other); University Hospital, Bordeaux (Other); University Hospital, Brest (Other); University Hospital, Lille (Other); University Hospital, Montpellier (Other); Saint Antoine University Hospital (Other); Pitié-Salpêtrière Hospital (Other); Hôpital Cochin (Other); Bicetre Hospital (Other); Bichat Hospital (Other); University Hospital, Rouen (Other); University Hospital, Strasbourg, France (Other); University Hospital, Toulouse (Other); University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: P030717
Record Dates: First submitted 2018-08-31; First posted 2018-09-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-07

CONDITIONS: Early Rheumatoid Arthritis or Early Undiffentiated Arthritis
Keywords: ESPOIR cohort RA Early Undifferentiated Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum at baseline, 6, 12, 18, 24, 36, 60, 120, 180 and 240 months / Urine at baseline, 24 and 36 months / DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The French Society of Rheumatology initiated a large national multicenter, longitudinal and prospective cohort, ESPOIR, in order to set up databases to allow various investigations on diagnosis, prognostic markers, epidemiology, pathogenesis and medico-economic factors in the field of early arthritis and rheumatoid arthritis.

The primary objective is to set-up a multicentre cohort of early arthritis (less than 6 months) in France that could serve as a database to studies of various natures.

Specific objectives are in the following domains:

* diagnosis: to help determine among clinical, biological, radiographic and immunogenetics those parameters allowing for the earliest diagnosis classification as possible, in order to target early therapy;
* prognosis: to identify early those patients at risk of severe disease by investigating among clinical, biological, genetic and sociologic factors;
* medico-economic: to identify the costs and their determinants at various disease stage;
* pathologic: to collect a databank of sera, DNA, RNA to allow for studies of transcriptomes and other genomics.

Secondary objectives are twofold:

* to monitor adverse events, particularly rare drug adverse events, in collaboration with other international studies
* to allow access to the data collected in this cohort study in order to facilitate new projects submitted to and approved by the scientific committee.

DETAILED DESCRIPTION:
All patients were referred to each regional center every 6 months during the first 2 years, then every year. Procedures were set up to avoid patients lost to followup as much as possible. At baseline and at each visit, we recorded data for a set of clinical and biological variables recommended for the management of early arthritis. At each visit, rheumatoid arthritis was classified according to the 1987 American College of Rheumatology (ACR) criteria and retrospectively to the 2010 ACR/European League Against Rheumatism (EULAR) criteria.

At each visit, patients completed function and quality-of-life self-administered questionnaires including the Health Assessment Questionnaire-Disability Index (HAQ-DI), Arthritis Impact Measurement Scales version 2 short form, a medico economic questionnaire, and globally assessed disease, pain at rest and pain during motion on a visual analog scale (VAS). Patients underwent radiographs of the hand and wrist (face) and foot (face and oblique). Radiographs were stored in the radiological coordinating center (Brest) and then were evaluated by the van der Heijde-modified Sharp score. Serum, DNA, urine, were collected at baseline. Serum and urine were also obtained at each follow-up visit. They were then sent and stored in adequate and definite conditions in the biological coordinating centre (Paris-Bichat).

ELIGIBILITY:
Inclusion Criteria:

* patients aged over 18 and under 70
* clinical diagnosis of rheumatoid arthritis as certain or probable
* clinical diagnosis of undifferentiated arthritis potentially becoming rheumatoid arthritis
* at least 2 inflammatory joints since 6 weeks : a swollen joint has to be observed in two articular sites and be present since at least 6 weeks
* arthritis starting since less than 6 months
* never prescribed DMARDS, corticoids, except if less than 2 weeks or except intra-articular injection less than 6 weeks before inclusion
* corticosteroids could be tolerated if prescribed for duration less than 2 weeks in the month before the inclusion with an average dose less than 20 mg per day and stopped two weeks before inclusion

Exclusion Criteria:

* patients aged less than 18 years or aged more than 70 years
* pregnant women
* undifferentiated rheumatism with no potential chance to become rheumatoid arthritis
* other inflammatory rheumatisms clearly defined

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 814 patients with early arthritis were included be- tween November 2002 and april 2005.One patient removed his consent form. All the centres were active and each regional centre recruited between 35 and 83 patients.
Sampling Method: Non-Probability Sample
Enrollment: 813 (Actual)
Dates: Start 2002-11-13 (Actual); Primary Completion 2005-04-19 (Actual); Study Completion 2025-07-13 (Actual)

PRIMARY OUTCOMES:
Remaining in the cohort. | 20 years
  Presence of the patient at the visit.
Prescription of synthetic or biologic disease-modifying antirheumatic drugs (DMARD). | 20 years
  Number of patients treated or not.
Patient disability evaluation. | 20 years
  Evaluation by Health Assessment Questionnaire Disability Index (HAQ-DI). The following categories are assessed by the HAQ-DI: dressing and grooming, arising, eating, walking, hygiene, reach, grip, common daily activities. The patients report the amount of difficulty they have in performing some of these activities. Each question asks on a scale ranging from 0 to 3. Increasing scores indicate worse functioning with 0 indicating no functional impairment and 3 indicating complete impairment.
Change in Disease Activity (levels of activity or remission) | 20 years
  1. Disease Activity Score (DAS28). The DAS28 provides an absolute indication of RA disease activity on a scale of 0.49 to 9.07 A DAS28 value >5.1 corresponds to a high disease activity, A DAS28 value between 3.2 and 5.1 corresponds to a moderate disease activity, A DAS28 value between 2.6 and 3.2 corresponds to a low disease activity, A DAS28 value < 2.6 corresponds to remission.
  2. Physician and patient activity VAS. Scales from 0 to 100. A high value indicates extreme activity.
Quality of life assessed by EQ-5D-3L/ EUROQOL | 20 years
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The EQ VAS records the respondent's self-rated health (0-100).
Quality of life assessed by MOS-SF-36/ MOS 36-Item Short-Form Health Survey | 15 years (from baseline to 15 years)
  MOS-SF-36/ MOS 36-Item Short-Form Health Survey contains 8 health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides the perceived change in health. Each dimension has a scale (0-100). Low score=poor quality of life.
Quality of life assessed by AIMS2-SF/Arthritis Impact Measurement Scales 2 Short Form | 14 years (from baseline to 14 years)
  AIMS2-SF/Arthritis Impact Measurement Scales 2 Short Form contains 26 items : upper-extremity functioning, lower-extremity functioning, affect, symptoms, social interaction, and role. Scores are summed and converted to a range of 0-10. Higher scores=poorer health.
Radiographic damage evaluation | 20 years
  Structural joint damage was assessed radiographically and expressed as change in Total Sharp Score (TSS) and its components.The SHS method evaluates, in each hand, 16 areas for erosions and 15 areas for JSN, and, in each foot, 6 areas for erosions and 6 areas for JSN. The erosion score per hand joint can range from 0 to 5. JSN and joint subluxation or luxation are combined in a single score, from 0 to 4. The maximal score for erosion and JSN are 160 and 120, respectively, for the hands and 120 and 48, respectively, for the feet. The maximal total SHS is 448.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard COMBE, MD, PHD, Principal Investigator — Montpellier University Hospital rheumatology department

REFERENCES:
- [Derived] Vittecoq O, Guillou C, Hardouin J, Gerard B, Berenbaum F, Constantin A, Rincheval N, Combe B, Lequerre T, Cosette P. Validation in the ESPOIR cohort of vitamin K-dependent protein S (PROS) as a potential biomarker capable of predicting response to the methotrexate/etanercept combination. Arthritis Res Ther. 2022 Mar 21;24(1):72. doi: 10.1186/s13075-022-02762-5. PMID 35313956
- [Derived] Kumaradev S, Roux C, Sellam J, Perrot S, Pham T, Dugravot A, Molto A. Socio-demographic determinants in the evolution of pain in inflammatory rheumatic diseases: results from ESPOIR and DESIR cohorts. Rheumatology (Oxford). 2022 Apr 11;61(4):1496-1509. doi: 10.1093/rheumatology/keab562. PMID 34270700
- [Derived] Roubille C, Coffy A, Rincheval N, Dougados M, Flipo RM, Daures JP, Combe B. Ten-year analysis of the risk of severe outcomes related to low-dose glucocorticoids in early rheumatoid arthritis. Rheumatology (Oxford). 2021 Aug 2;60(8):3738-3746. doi: 10.1093/rheumatology/keaa850. PMID 33320245
- [Derived] Valdeyron C, Soubrier M, Pereira B, Constantin A, Morel J, Gaudin P, Combe B, Gremeau AS, Dejou-Bouillet L, Pouly JL, Sapin V, Oris C, Brugnon F. Impact of disease activity and treatments on ovarian reserve in patients with rheumatoid arthritis in the ESPOIR cohort. Rheumatology (Oxford). 2021 Apr 6;60(4):1863-1870. doi: 10.1093/rheumatology/keaa535. PMID 33147613
- [Derived] Mouterde G, Gamon E, Rincheval N, Lukas C, Seror R, Berenbaum F, Dupuy AM, Daien C, Daures JP, Combe B. Association Between Vitamin D Deficiency and Disease Activity, Disability, and Radiographic Progression in Early Rheumatoid Arthritis: The ESPOIR Cohort. J Rheumatol. 2020 Nov 1;47(11):1624-1628. doi: 10.3899/jrheum.190795. Epub 2019 Dec 15. PMID 31839594
- [Derived] Lukas C, Mary J, Debandt M, Daien C, Morel J, Cantagrel A, Fautrel B, Combe B. Predictors of good response to conventional synthetic DMARDs in early seronegative rheumatoid arthritis: data from the ESPOIR cohort. Arthritis Res Ther. 2019 Nov 15;21(1):243. doi: 10.1186/s13075-019-2020-x. PMID 31730497